CLINICAL TRIAL: NCT01963468
Title: Pre-Implantation Communication Treatment for Children With Hearing Loss
Brief Title: Maximizing Language Development in Children With Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Megan Roberts, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00081066; 1R03DC012639 (NIH)
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Hearing Loss
Keywords: Hearing Loss; Cochlear Implant; Deaf; Hearing Impairment; Hard of Hearing
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early language intervention (Experimental): Children will receive 6 months of weekly parent-implemented intervention sessions.
  Children will be assessed monthly via audio recordings and language checklists to monitor language development more closely.
  Interventions: Behavioral: Early language intervention
- Monthly language check-ups (No Intervention): Children will be assessed monthly via home observations and parents will complete a language checklist to monitor language development more closely.

INTERVENTIONS:
Behavioral: Early language intervention — Parents will practice the specific set of strategies (visual, interactive, tactile, responsive) during sessions that occur weekly and last 1 hour for a total of 26 sessions, over 6 months. Each session will include four segments: (a) the therapist will review the intervention strategies taught in the workshop (10 min), (b) the therapist will model the intervention strategy with the child (10 min), (c) the parent will practice the strategy with her child with coaching from the therapist across four different routines and activities of the parent's choice (30 min), and (d) the therapist will provide feedback to the parent, summarize the session, and answer the parent's questions (10 min).
  Arms: Early language intervention

SUMMARY:
The purpose of this study is to evaluate the effects of early intervention on language skills for children with hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 18 months of age
* bilateral, moderate to profound congenital hearing loss

Exclusion Criteria:

* auditory neuropathy
* no known additional disabilities (e.g., cerebral palsy, Down syndrome)
* both parents have a severe to profound hearing loss

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
MacArthur Communicative Development Inventories | one month

SECONDARY OUTCOMES:
Preschool Language Scale | 6 months

OTHER OUTCOMES:
Communication and Symbolic Behavior Scales | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Megan Y Roberts, PhD, CCC-SLP, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Evanston, Illinois, United States